CLINICAL TRIAL: NCT00576108
Title: A 2 Week Study of Topical KD7040 in the Treatment of Postherpetic Neuralgia (PHN)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kalypsys, Inc. (Industry)
Responsible Party: Kalypsys, Inc., Kalypsys, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KD7040-NP02
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Postherpetic Neuralgia; Shingles; Herpes Zoster; Neuropathic Pain
MeSH Terms: conditions — Neuralgia, Postherpetic; Herpes Zoster; Neuralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- KD7040 topical gel (Experimental)
  Interventions: Drug: KD7040 Topical Gel
- Placebo gel (Placebo Comparator)
  Interventions: Drug: Placebo gel

INTERVENTIONS:
Drug: KD7040 Topical Gel — KD7040 topical gel
  Arms: KD7040 topical gel
Drug: Placebo gel — Placebo gel
  Arms: Placebo gel

SUMMARY:
This study will evaluate the safety and efficacy of 2 weeks of topical KD7040 versus placebo in the treatment of postherpetic neuralgia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ages 18-85 years
* Previous diagnosis of Shingles (Herpes Zoster) with pain persisting for at least 3 months, but not longer than 5 years, after healing of rash
* Subject with intact skin in the targeted treatment area
* Female subjects of childbearing potential must have a negative serum pregnancy test at screening, a negative urine human chorionic gonadotropin (hCG) test prior to randomization, and must use medically acceptable methods of birth control. All subjects must agree to take every precaution to ensure that pregnancy will not occur during the study.
* Subject must be willing and able to complete screening and study procedures as described int he protocol.
* Subject must voluntarily provide written Informed Consent prior to participation.

Exclusion Criteria:

* Subjects with known hypersensitivity to KD7040 or methylparaben, or previous exposure to KD7040.
* Subjects pregnant, nursing or planning to become pregnant.
* Subjects who are immunocompromised or have clinically significant hematological abnormalities.
* Subjects with system dermatological conditions (e.g., psoriasis, atopic dermatitis) or impaired wound healing.
* Subjects who have had local anesthetic nerve blocks within 48 hours of study entry.
* Subjects having other sever pain which may confound assessment of PHN.
* Subjects who have serious, unstable, or clinically significant medical or psychological conditions, which, in the opinion of the Investigator(s) would compromise the subjects' participation in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Worst daily pain | Once daily

SECONDARY OUTCOMES:
Average daily pain | Once daily

CONTACTS AND LOCATIONS:
Locations (1):
- United Bioscience Corporation, Kansas City, Missouri, United States